CLINICAL TRIAL: NCT06003114
Title: Real-World Utilization of Palbociclib as 1L Treatment in Canadian HR+/HER2-women Breast Cancer Patients
Brief Title: A Study to Understand the Use of Palbociclib in Canadian Patients With Breast Cancer That Has Spread to Other Organs
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5481183; PALCAN (Other: Alias Study Number)
Record Dates: First submitted 2023-08-10; First posted 2023-08-21 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer
Keywords: Metastatic breast cancer (MBC); Human epidermal growth factor receptor 2 negative (HER2-); Hormone receptor positive (HR+); First line; Real world
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- First-line patients on Palbociclib: Participants taking oral palbociclib as prescribed in first-line treatment
  Interventions: Drug: Palbociclib

INTERVENTIONS:
Drug: Palbociclib — Participants taking oral palbociclib as prescribed in first-line treatment.
  Other Names: Ibrance

SUMMARY:
The purpose of this real-world study is to understand the use of palbociclib as first treatment for Hormone receptor positive (HR+) and Human epidermal growth factor receptor 2 negative (HER2-) metastatic breast cancer in Canada (PALCAN).

The real-world study is not a research study. It involves real patients who receive medicines prescribed by their doctors in the real world. Metastatic breast cancer is the type which has spread from breast to other organs.

HR positive stands for Hormone-receptor cells that have a protein on their surface that binds to one of 2 types of hormones. They are estrogen or progesterone. Both these hormones help cancer cells grow.

HER2 negative describes cells that have a small amount or none of a protein called HER2 on their surface. In normal cells, HER2 helps control cell growth. Cancer cells that are HER2 negative may grow more slowly and are less likely to come back or spread to other parts of the body.

This study will mainly measure:

- duration of treatment (from start of treatment till end of treatment) among a group of patients taking palbociclib (Ibrance) in combination with hormone therapy as first line treatment for HR+ HER2- metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Received at least one cycle of palbociclib as first line therapy for metastatic breast cancer between 01 January 2016 and 31 December 2022
* Histologically confirmed HR+/HER2- metastatic breast cancer
* Minimum of 3 months available follow-up on palbociclib

Exclusion Criteria:

* Received a different CDK4/6 inhibitor before palbociclib in the first line
* Received other systemic therapy, including hormone therapy, 15-60 days prior to initiation of palbociclib
* Invalid or incomplete records (more specifically, complete duration of treatment on palbociclib, endocrine therapy or LHRH)
* Death date recorded on or before the date of index date

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Treatment of Canadian women patients on palbociclib with HR+/HER2- metastatic breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 472 (Actual)
Dates: Start 2023-10-06 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
Estimate the median Duration of Treatment (DoT) | Time index of approximately 01 Jan 2016 to 31 March 2022

SECONDARY OUTCOMES:
Number of patients with treatment discontinuation at one-year intervals | Time index of approximately 01 Jan 2016 to 31 March 2022
Number of patients starting at initial dose | Time index of approximately 01 Jan 2016 to 31 March 2022
Time to chemotherapy | Time index of approximately 01 Jan 2016 to 31 March 2022
Clinical Characteristics of Patients | Time index of approximately 01 Jan 2016 to 31 March 2022
Demographical Characteristics of Patients | Time index of approximately 01 Jan 2016 to 31 March 2022

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Alberta Health Services, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A5481183